CLINICAL TRIAL: NCT04067440
Title: Characterization and Comparison of the Human Microbiome in Peritoneum, Jejunum, Rectum and Stool
Brief Title: Characterization of the Microbiome in Peritoneum, Jejunum, Rectum and Stool
Acronym: METABIOM
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Michael Jelden, Dr. med. Michael Jelden, University Hospital, Saarland
Other Study IDs: METABIOM
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Diabetes Mellitus; Fatty Liver, Nonalcoholic; Leaky Gut Syndrome; Chronic Pancreatitis
Keywords: Microbiome; Obesity; Chronic Liver Disease
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Subjects to undergo surgery including opening of the jejunum with non-inflammative condition.
  Interventions: Diagnostic Test: Microbial Swab

INTERVENTIONS:
Diagnostic Test: Microbial Swab — Swabs will be taken from peritoneum and jejunum (intraoperatively), rectum, and stool

SUMMARY:
Characterization of the human microbiome in the jejunum and comparison to the microbiome in the rectum and stool in order to see how the microbial communities change within the intestines.

DETAILED DESCRIPTION:
Subjects to undergo surgery with opening of the jejunum will be sampled with sterile swabs from peritoneum and the inside of the jejunum. A swab will also be taken from the rectum.

The peritoneum is regarded as a sterile place until today. We try to either verify this, we also could find a scientific base for theories like leaky gut or other forms of bacterial migration through the intestinal wall.

Many of these patients undergo bariatric surgery. Many of them do have a dramatic change in glucose metabolism immediate after surgery. Therefore stool swabs will be taken before and 5 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* abdominal surgery containing opening of jejunum
* singing of consent

Exclusion Criteria:

* inflammative condition (appendicitis, pancreatitis, Crohn, Colitis ulcerous, cholecystitis and similar)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obesity
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Characterization of microbiome | intra-operative
  Previously uncharacterized sites: jejunum, peritoneum

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jelden, Dr., Principal Investigator — Saarland University Hospital
Locations (1):
- Department of General, Visceral, Vascular and Pediatric Surgery, University of Saarland,, Homburg/Saar, Germany

IPD SHARING:
Plan to Share IPD: Undecided